CLINICAL TRIAL: NCT00552032
Title: A Double-blind Placebo-controlled, Randomized, Parallel-group, Multicenter Clinical Trial to Evaluate Efficacy and Safety of Mometasone Furoate Nasal Spray in Children With Adenoid Hypertrophy SNORE Study
Brief Title: Efficacy and Safety of Mometasone Furoate Nasal Spray in Children With Adenoid Hypertrophy. SNORE Study (P05155)
Acronym: SNORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05155
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2012-01-31 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Adenoids Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone Furoate nasal spray (Experimental)
  Interventions: Drug: Mometasone Furoate nasal spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate nasal spray — Mometasone Furoate nasal spray 1 puff (50 mcg) per nostril twice daily x 8 weeks. There was a blinded follow-up period of 16 weeks, resulting in study duration of 24 weeks (6 months).
  Other Names: SCH 032088
  Arms: Mometasone Furoate nasal spray
Drug: Placebo — Placebo nasal spray 1 puff per nostril twice daily x 8 weeks. There was a blinded follow-up period of 16 weeks, resulting in study duration of 24 weeks (6 months).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether 8 weeks treatment with mometasone furoate nasal spray (MFNS), twice daily, is safe and effective in treating adenoid hypertrophy in children.

ELIGIBILITY:
Inclusion Criteria:

* Participants and their parents must demonstrate willingness to participate and comply with study procedures. Parents must sign a written informed consent
* Participants and their parents must understand and be able to adhere to dosing and visit schedules, and agree to record symptom severity scores, medication times, and concomitant medications accurately and consistently in a daily diary
* Children with a history of adenoid hypertrophy for at least 3 months with no response to previous medical treatment
* Baseline adenoid tissue size must have been graded by nasopharyngoscopy examination as Grade III or IV on the Adenoid/Choana (A/C) Index (between 50% and 100% obstruction)
* Baseline Total Severity Symptoms Score must be ≥ 8 points (AM or PM)
* For inclusion in endpoints relating to otitis media with effusion (OME), participant must have persistent middle ear effusion for the past 3 months or more documented by otoscopic examination, middle ear pressure less than -150 mm H2O, Jerger type B flat tympanogram, and mild-moderate conductive hearing loss in audiometry supporting the diagnosis of OME

Exclusion Criteria:

* Participants with previous surgery of hypertrophic adenoids with or without tympanostomy tube placement
* Participants treated with inhaled or systemic corticosteroids within the past 1 month
* Participants with Morbid Obesity (Body Mass Index >95 percentile of charts from the Centers for Disease Control)
* Participants who have not accomplished the designated washout periods for any of the prohibited medications
* Participants who have used any investigational products within the last 30 days
* Participants who have used any antibodies for allergies in the past 90 days
* Participants who have any abnormal physical examination results that may affect study evaluations or participant safety in the investigator's judgment
* Participants who are allergic or have an idiosyncratic reaction to corticosteroids
* Participants with signs and symptoms of acute or chronic bacterial rhinosinusitis
* Participants has had an upper or lower respiratory tract or sinus infection that required antibiotic therapy with the last dose later than 14 days prior to screening, or who has had a viral upper or lower respiratory infection within 7 days prior to screening
* Participants with a documented immunodeficiency condition
* Participants with nasal structural abnormalities, including large nasal polyps and marked septum deviation that significantly interferes with nasal airflow
* Participants with any clinically significant metabolic, cardiovascular, neurologic, hematologic, gastrointestinal, cerebrovascular, or respiratory disease (other than asthma), or any other disorder which, in the judgment of the Investigator, may interfere with the study evaluations or affect participant safety

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-01-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 135 participants were screened, a total of 132 participants were randomized to receive either Mometasone furoate nasal spray (MFNS) (n=66) or placebo nasal spray (n=66).
Groups:
- Mometasone Furoate Nasal Spray: 1 spray (50 mcg) in each nostril twice daily (equivalent to 200 mcg per day) administered for 8 weeks. There was a blinded follow-up period of 16 weeks, resulting in study duration of 24 weeks (6 months).
- Placebo Nasal Spray: 1 spray in each nostril twice daily administered for 8 weeks. There was a blinded follow-up period of 16 weeks, resulting in study duration of 24 weeks (6 months).
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Started | 66 | 66
Completed | 49 | 47
Not Completed | 17 | 19
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 7 | 12
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.56 (2.27) | 5.36 (2.50) | 5.46 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 23 | 55
  Male | 34 | 43 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adenoid/Choana (A/C) Index Grade
Description: Changes in adenoid size were assessed by nasopharyngoscopic examination and were determined using the Adenoid/Choana (A/C) Index. Grades were assigned to intervals of A/C ratio percentages: grade I (0-25%), II (26-50%), III (51-75%) and IV (76-100%). Changes in adenoid size were expressed as the mean difference between grades at baseline and study visit. Positive values indicated a decrease in adenoid size, a 0 value indicated that size remained the same, and negative values indicated an increase in adenoid size.
Time Frame: Baseline (visit 2), Weeks 4 (visit 3), Week 8 (visit 4)
Population: A total of 132 participants were included in the intent-to-treat (ITT) population. The ITT population included all randomized participants who received at least one dose after commencement of treatment. Data are summarized in terms of the number of participants providing data at the relevant time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Mometasone Furoate Nasal Spray (MFNS): 1 spray (50 mcg) in each nostril twice daily (equivalent to 200 mcg per day) administered for 8 weeks. There was a blinded follow-up period of 16 weeks, resulting in study duration of 24 weeks (6 months).
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Score on a Scale
  Change at Visit 3 (n=65 MFNS, n=63 Placebo) | 0.3 (0.6) | 0.2 (0.5)
  Change at Visit 4 (n=61 MFNS, n=58 Placebo) | 0.4 (0.7) | 0.3 (0.7)

2. Secondary Outcome: Total Severity Symptom Scores: Morning and Evening (AM & PM)
Description: Symptoms were assessed by whole-number linear scale to grade their severity. Scores were recorded AM & PM (a difference of 12 hours) & were based on severity within 12 hours of prior recording. The following symptoms were evaluated: Snoring; Nasal obstruction & discharge; Breathing difficulty; Oral respiration; Ear pain. Severity was graded according to the following scale: 0=absent; 1=mild; 2=moderate; 3=severe. Severity was scored individually and summed to obtain the Total Symptom Severity Score. The maximum total score possible was 36 daily; 18 for both AM (6 symptoms times max severity of 3)and PM.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: A total of 132 participants were included in the ITT population. The ITT population included all randomized participants who received at least one dose after commencement of treatment. Data summarized in terms of the number of participants providing data at the relevant time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Score on a scale
  Visit 2 AM (n=66 MFNS, n=66 Placebo) | 9.4 (2.5) | 9.9 (3.3)
  Visit 3 AM (n=64 MFNS, n=65 Placebo) | 5.4 (3.8) | 6.4 (3.7)
  Visit 4 AM (n=62 MFNS, n=60 Placebo) | 4.2 (3.6) | 5.5 (3.5)
  Visit 2 PM (n=66 MFNS, n=66 Placebo) | 9.9 (3.2) | 10.2 (2.8)
  Visit 3 PM (n=64 MFNS, n=65 Placebo) | 6.3 (3.7) | 7.0 (3.6)
  Visit 4 PM (n=62 MFNS, n=60 Placebo) | 4.8 (3.8) | 5.7 (3.8)

3. Secondary Outcome: Total Frequency Symptom Scores: AM & PM
Description: Symptoms were assessed by whole-number linear scale to grade their frequency. Scores were recorded AM & PM (a difference of 12 hours) & were based on frequency within 12 hours of prior recording. The following signs/symptoms were evaluated: Snoring; Nasal obstruction; and nasal discharge; Breathing difficulty; Oral respiration; Ear pain. Frequency was graded according to the following scale: 0=absent; 1=intermittent; 2=persistent. The frequency of symptoms was scored individually and summed to obtain the Total Frequency Symptom Score. The maximum total score possible was 24 daily; 12 for both AM (6 symptoms times max frequency of 2) and PM.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Score on a scale
  Visit 2 AM (n=66 MFNS, n=66 Placebo) | 7.3 (1.9) | 7.3 (2.4)
  Visit 3 AM (n=64 MFNS, n=65 Placebo) | 4.4 (2.7) | 5.4 (2.6)
  Visit 4 AM (n=62 MFNS, n=60 Placebo) | 3.7 (2.8) | 4.4 (2.5)
  Visit 2 PM (n=66 MFNS, n=66 Placebo) | 7.6 (2.2) | 8.0 (2.1)
  Visit 3 PM (n=64 MFNS, n=65 Placebo) | 5.3 (2.8) | 5.7 (2.6)
  Visit 4 PM (n=62 MFNS, n=60 Placebo) | 4.1 (2.9) | 4.6 (2.7)

4. Secondary Outcome: Number of Participants With Bilateral Tympanogram Results of: Normal, Abnormal, or Not Done
Description: Tympanometry was performed in children ages 2-11 by certified audiologists. Results were categorized based on audiologist's assessment as either being normal (normal pressure in the middle ear with normal mobility of the eardrum and the conduction bones) , abnormal (abnormal pressure in the middle ear and/or abnormal mobility of the eardrum and the conduction bones), or tympanometry was not done (evaluation not completed). Results were assessed at baseline, Week 4 (Visit 3), and endpoint Week 8 (end of treatment).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Participants
  Visit 2- Normal (n=66 MFNS, n=66 Placebo) | 35 | 39
  Visit 2- Abnormal (n=66 MFNS, n=66 Placebo) | 25 | 22
  Visit 2- Not Done (n=66 MFNS, n=66 Placebo) | 6 | 5
  Visit 3- Normal (n=65 MFNS, n=65 Placebo) | 44 | 33
  Visit 3- Abnormal (n=65 MFNS, n=65 Placebo) | 14 | 22
  Visit 3- Not Done (n=65 MFNS, n=65 Placebo) | 7 | 10
  Visit 4- Normal (n=62 MFNS, n=60 Placebo) | 45 | 39
  Visit 4- Abnormal (n=62 MFNS, n=60 Placebo) | 16 | 19
  Visit 4- Not Done (n=62 MFNS, n=60 Placebo) | 1 | 2

5. Secondary Outcome: Number of Participants With Otoscopic Results of: Normal or Abnormal
Description: Otoscopic examination was performed of the right and left ear canals at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4). Results were categorized based on audiologist's assessment as either being normal (ear canal structures appear normal) or abnormal (ear canal structures appear abnormal).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Participants
  Right Otoscopy: Visit 2- Normal (n=66, n=66) | 50 | 51
  Right Otoscopy: Visit 2- Abnormal (n=66, n=66) | 16 | 15
  Right Otoscopy Visit 3- Normal (n=65, n=65) | 54 | 53
  Right Otoscopy Visit 3- Abnormal (n=65, n=65) | 11 | 12
  Right Otoscopy Visit 4- Normal (n=62, n=60) | 49 | 52
  Right Otoscopy Visit 4- Abnormal (n=62, n=60) | 13 | 8
  Left Otoscopy: Visit 2- Normal (n=66, n=66) | 49 | 52
  Left Otoscopy: Visit 2- Abnormal (n=66, n=66) | 17 | 14
  Left Otoscopy Visit 3- Normal (n=65, n=65) | 51 | 55
  Left Otoscopy Visit 3- Abnormal (n=65, n=65) | 14 | 10
  Left Otoscopy Visit 4- Normal (n=62, n=60) | 48 | 52
  Left Otoscopy Visit 4- Abnormal (n=62, n=60) | 14 | 8

6. Secondary Outcome: Number of Participants With Rhinoscopic- Septum Results of: Aligned, Non-Obstructive, or Obstructive Deviation
Description: Rhinoscopic examination of the septum was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4). Results were categorized based on investigator's assessment as either being aligned (septum is aligned), non-obstructive (septum is not aligned but the deviation is non-obstructive), or obstructive (septum is deviated and obstructive) deviation.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Participants
  Visit 2 Aligned (n= 66, n=66) | 65 | 63
  Visit 2 Non-obstructive Deviation (n= 66, n=66) | 1 | 3
  Vist 2 Obstructive Deviation (n=66, n=66) | 0 | 0
  Visit 3 Aligned (n=65, n=65) | 64 | 62
  Visit 3 Non-obstructive Deviation (n=65, n=65) | 1 | 3
  Visit 3 Obstructive Deviation (n=65, n=65) | 0 | 0
  Visit 4 Aligned (n=62, n=60) | 61 | 57
  Visit 4 Non-obstructive Deviation (n=62, n=60) | 1 | 3
  Visit 4 -Obstructive Deviation (n=62, n=60) | 0 | 0

7. Secondary Outcome: Number of Participants With Rhinoscopic-Inferior Turbinates Results of: Normal, Hypertrophic, and Hypotrophic
Description: Rhinoscopic examination of the inferior turbinates was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4). Results were categorized based on investigator's assessment as either being normal appearance (normal size) , hypertrophic (swollen/normal size increased), or hypotrophic (normal size diminished).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Participants
  Visit 2- Normal Appearance (n=66, n=66) | 50 | 46
  Visit 2 Hypertrophic (n=66, n=66) | 16 | 20
  Vist 2 Hypotrophic (n=66, n=66) | 0 | 0
  Visit 3 Normal Appearance (n=65, n=65) | 46 | 48
  Visit 3 Hypertrophic (n=65, n=65) | 19 | 17
  Visit 3 Hypotrophic (n=65, n=65) | 0 | 0
  Visit 4 Normal Appearance (n=62, n=60) | 45 | 42
  Visit 4 Hypertrophic (n=62, n=60) | 17 | 18
  Visit 4 Hypotrophic (n=62, n=60) | 0 | 0

8. Secondary Outcome: Number of Participants With Rhinoscopic- Middle Meatus Results of: Patent, Partial Obstruction or Total Obstruction
Description: Rhinoscopic examination of the middle meatus was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4). Results were categorized based on investigator's assessment into 3 categories: patent (easily observed), partial obstruction (partially blocked from view), or total obstruction (completely blocked from view).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Participants
  Visit 2- Patent (n=66, n=66) | 62 | 60
  Visit 2- Partial Obstruction (n=66, n=66) | 3 | 5
  Visit 2- Total Obstruction (n=66, n=66) | 1 | 1
  Visit 3- Patent (n=65, n=65) | 61 | 61
  Visit 3- Partial Obstruction (n=65, n=65) | 4 | 2
  Visit 3- Total Obstruction (n=65, n=65) | 0 | 2
  Visit 4- Patent (n=62, n=60) | 56 | 53
  Visit 4- Partial Obstruction (n= 62, n=60) | 6 | 4
  Visit 4- Total Obstruction (n=62, n=60) | 0 | 3

9. Secondary Outcome: Rhinomanometry Results- Left and Right Nasal Fossa: Inspiratory Resistance
Description: Rhinomanometry examination of the left & right Nasal Fossa was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4) in participants ages 7-11 years.
  Rhinomanometry is a test of nasal function that measures air pressure and the rate of airflow in the nasal airway during respiration by means of equipment. These findings were used to calculate inspiratory nasal airway resistance reported in Pascal/centimeter^3/second (Pa/cm^3/sec).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants aged 7-11 years old (MFSN=19, Placebo=20).
Measure: Mean (Standard Deviation); unit: Pa/cm^3/sec
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
Pa/cm^3/sec
  Visit 2- Left Nasal Fossa (n=19, n=20) | 2.111 (4.372) | 3.280 (7.852)
  Visit 3- Left Nasal Fossa (n=18, n=18) | 6.341 (22.759) | 1.934 (2.234)
  Visit 4- Left Nasal Fossa (n=19, n=19) | 31.074 (131.718) | 54.724 (229.437)
  Visit 2- Right Nasal Fossa (n=19, n=20) | 2.985 (8.527) | 6.535 (24.836)
  Visit 3- Right Nasal Fossa (n=18, n=18) | 1.823 (4.454) | 3.026 (8.258)
  Visit 4- Right Nasal Fossa (n=19, n=19) | 2.560 (6.918) | 43.621 (174.535)

10. Secondary Outcome: Rhinomanometry Results- Left and Right Nasal Fossa: Expiratory Resistance
Description: Rhinomanometry examination of the left & right Nasal Fossa was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4) in participants ages 7-11 years.
  Rhinomanometry is a test of nasal function that measures air pressure and the rate of airflow in the nasal airway during respiration by means of equipment. These findings were used to calculate expiratory nasal airway resistance reported in Pascal/centimeter^3/second (Pa/cm^3/sec).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants ages 7-11 years old (MFSN=19, Placebo=20).
Measure: Mean (Standard Deviation); unit: Pa/cm^3/sec
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
Pa/cm^3/sec
  Visit 2- Left Nasal Fossa (n=19, n=20) | 1.771 (2.764) | 3.994 (9.416)
  Visit 3- Left Nasal Fossa (n=18, n=18) | 2.937 (8.196) | 1.478 (1.647)
  Visit 4- Left Nasal Fossa (n=19, n=19) | 13.488 (32.344) | 4.148 (13.999)
  Visit 2- Right Nasal Fossa (n=19, n=20) | 2.625 (6.868) | 1.083 (1.109)
  Visit 3- Right Nasal Fossa (n=18, n=18) | 2.189 (4.678) | 3.646 (8.313)
  Visit 4- Right Nasal Fossa (n=19, n=19) | 0.961 (0.758) | 2.792 (6.318)

11. Secondary Outcome: Rhinomanometry Results- Left and Right Nasal Fossa: Inspiration Flow at 75 Pa
Description: Rhinomanometry examination of the left & right Nasal Fossa was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4) in participants ages 7-11 years.
  Rhinomanometry is a test of nasal function that measures air pressure and the rate of airflow in the nasal airway during respiration by means of equipment. Inspiration flow was calculated at 75 Pa.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants ages 7-11 years old (MFSN=19, Placebo=20).
Measure: Mean (Standard Deviation); unit: cm^3/sec
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
cm^3/sec
  Visit 2- Left Nasal Fossa (n=19, n=20) | 200.530 (140.492) | 178.933 (129.272)
  Visit 3- Left Nasal Fossa (n=18, n=18) | 222.152 (141.740) | 151.268 (130.115)
  Visit 4- Left Nasal Fossa (n=19, n=19) | 194.208 (100.746) | 172.346 (102.607)
  Visit 2- Right Nasal Fossa (n=19, n=20) | 183.562 (121.780) | 161.958 (138.673)
  Visit 3- Right Nasal Fossa (n=18, n=18) | 228.661 (149.318) | 197.266 (123.763)
  Visit 4- Right Nasal Fossa (n=19, n=19) | 215.400 (157.794) | 183.368 (117.677)

12. Secondary Outcome: Rhinomanometry Results- Left and Right Nasal Fossa: Expiratory Flow at 75 Pa
Description: Rhinomanometry examination of the left & right Nasal Fossa was performed at baseline (visit 2) and each visit throughout treatment (visit 3 and visit 4) in participants ages 7-11 years.
  Rhinomanometry is a test of nasal function that measures air pressure and the rate of airflow in the nasal airway during respiration by means of equipment. Expiratory flow was calculated at 75 Pa.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants ages 7-11 years old (MFSN=19, Placebo=20).
Measure: Mean (Standard Deviation); unit: cm^3/sec
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
cm^3/sec
  Visit 2- Left Nasal Fossa (n=19, n=20) | 190.024 (146.067) | 166.930 (116.802)
  Visit 3- Left Nasal Fossa (n=18, n=18) | 225.911 (154.830) | 173.139 (151.783)
  Visit 4- Left Nasal Fossa (n=19, n=19) | 181.026 (119.728) | 192.374 (134.337)
  Visit 2- Right Nasal Fossa (n=19, n=20) | 160.531 (117.988) | 166.302 (132.754)
  Visit 3- Right Nasal Fossa (n=18, n=18) | 209.676 (157.215) | 209.787 (151.298)
  Visit 4- Right Nasal Fossa (n=19, n=19) | 195.108 (163.411) | 176.587 (111.421)

13. Secondary Outcome: Number of Participants With Pure-Tone Audiometric Results of: Normal, Abnormal, or Not Done
Description: Pure-tone audiometry was performed in children ages 7-11 by certified audiologists. Results were categorized based on audiologist's assessment as either being normal (within normal limits), abnormal (outside normal limits), or audiometry was not done (not performed). Results were assessed at baseline, Week 4 (Visit 3), and endpoint Week 8 (end of treatment).
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants ages 7-11 years old (MFSN=19, Placebo=20).
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
Participants
  Visit 2- Normal (n=19 MFNS, n=21 Placebo) | 13 | 18
  Visit 2- Abnormal (n=19 MFNS, n=21 Placebo) | 5 | 2
  Visit 2- Not Done (n=19 MFNS, n= 21 Placebo) | 1 | 1
  Visit 3- Normal (n=20 MFNS, n=21 Placebo) | 15 | 20
  Visit 3- Abnormal (n=20 MFNS, n=21 Placebo) | 4 | 1
  Visit 3- Not Done (n=20 MFNS, n=21 Placebo) | 1 | 0
  Visit 4- Normal (n=19 MFNS, n=20 Placebo) | 15 | 18
  Visit 4- Abnormal (n=19 MFNS, n=20 Placebo) | 2 | 2
  Visit 4- Not Done (n=19 MFNS, n=20 Placebo) | 2 | 0

14. Secondary Outcome: Acoustic Rhinometry Results- Minimal Cross-Sectional Area: Left and Right Nasal Fossa
Description: Acoustic rhinometry examination of the left & right Nasal Fossa was performed by principal investigators at baseline & each visit throughout treatment in participants ages 7-11 years. Acoustic rhinometry is a technique intended for assessment of the geometry of the nasal cavity and nasopharynx and for evaluating nasal obstruction. The technique is based on an analysis of sound waves reflected from the nasal cavities.
  Measurements were taken for each side of the nose (nasopharyngeal minimum cross-sectional area) & were reported in cm^3.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants ages 7-11 years old (MFSN=19, Placebo=20).
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
cm^3
  Visit 2- Left Nasal Fossa (n=19, n=20) | 0.599 (0.567) | 0.491 (0.265)
  Visit 3- Left Nasal Fossa (n=18, n=18) | 0.608 (0.485) | 0.594 (0.403)
  Visit 4- Left Nasal Fossa (n=19, n=19) | 0.662 (0.444) | 0.661 (0.444)
  Visit 2- Right Nasal Fossa (n=19, n=20) | 0.532 (0.467) | 0.577 (0.381)
  Visit 3- Right Nasal Fossa (n=18, n=18) | 0.581 (0.405) | 0.596 (0.383)
  Visit 4- Right Nasal Fossa (n=19, n=19) | 0.734 (0.599) | 0.814 (0.675)

15. Secondary Outcome: Acoustic Rhinometry Results- Nasopharyngeal Volume (NPV): Left and Right Nasal Fossa
Description: Acoustic rhinometry examination of the left & right Nasal Fossa was performed by principal investigators at baseline & each visit throughout treatment in participants ages 7-11 years. Acoustic rhinometry is a technique intended for assessment of the geometry of the nasal cavity and nasopharynx and for evaluating nasal obstruction. The technique is based on an analysis of sound waves reflected from the nasal cavities.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: This analysis was only performed in a cohort of the ITT in participants ages 7-11 years old (MFSN=19, Placebo=20).
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 19 | 20
cm^3
  Visit 2- Left Nasal Fossa (n=19, n=20) | 4.245 (1.954) | 4.117 (3.554)
  Visit 3- Left Nasal Fossa (n=18, n=18) | 3.725 (1.944) | 3.489 (1.589)
  Visit 4- Left Nasal Fossa (n=19, n=19) | 3.631 (0.905) | 3.084 (1.724)
  Visit 2- Right Nasal Fossa (n=19, n=20) | 3.566 (1.629) | 4.489 (2.941)
  Visit 3- Right Nasal Fossa (n=19, n=18) | 4.183 (1.341) | 4.884 (3.591)
  Visit 4- Right Nasal Fossa (n=19, n=19) | 3.774 (1.240) | 3.275 (1.083)

16. Secondary Outcome: Number of Participants With Pediatric Sleep Questionnaire (PSQ)- Impact on Health-Related Quality of Life (HRQL) Results of: Mild, Moderate, or Severe
Description: PSQ consists of 90 variables divided into 3 different factors:snoring, somnolence, and behavior. All positive Snoring and Somnolence answers scored with Yes=1 and No=0, and scores averaged to obtain a total score between 0.00 and 1.00. Behavior factor scored between 1-3, and scores averaged for total score of 1 to 3. Increased scores indicate increasing abnormality of sleep. Based on determined cut-offs, participants were categorized as having mild, moderate, or severe discomfort due to interference of sleep.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 65
Participants
  Visit 2- Mild (n=66 MFNS, n=65 Placebo) | 33 | 30
  Visit 2- Moderate (n=66 MFNS, n=65 Placebo) | 17 | 26
  Visit 2- Severe (n=66 MFNS, n=65 Placebo) | 16 | 9
  Visit 3- Mild (n=65 MFNS, n=65 Placebo) | 50 | 45
  Visit 3- Moderate (n=65 MFNS, n=Placebo) | 11 | 17
  Visit 3- Severe (n=65 MFNS, n=65 Placebo) | 4 | 3
  Visit 4- Mild (n=62 MFNS, n=59 Placebo) | 49 | 47
  Visit 4- Moderate (n=62 MFNS, n=59 Placebo) | 13 | 10
  Visit 4- Severe (n=62 MFNS, n= 59 Placebo) | 0 | 2

17. Secondary Outcome: Quality of Life Questionnaire (PedsQL) Total Score (Ages 2-4)
Description: The impact on quality of life (QOL) was measured by a general pediatric health questionnaire. Versions were self-administered & answered by participants' parents. This modular instrument consists of 21 items using a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored. Total score is sum of all the items over the number of items answered on all the scales. Higher scores indicate a better health related QOL.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: The ITT population included all randomized participants who received >= 1 dose after commencement of treatment. At baseline (visit 2), 52 randomized participants were between 2 and 4 years old, 23 participants in MFNS & 29 participants in Placebo group. Questionnaire was answered in accordance with the actual age of each participant at each visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 23 | 29
Score on a scale
  Visit 2 (n= 23 MFNS, n=29 Placebo) | 78.442 (13.114) | 78.017 (14.769)
  Visit 3 (n=22 MFNS, n= 28 Placebo) | 80.438 (15.827) | 78.486 (15.707)
  Visit 4 (n=18 MFNS, n=25 Placebo) | 80.137 (15.161) | 82.701 (11.911)

18. Secondary Outcome: Quality of Life Questionnaire (PedsQL) Total Score (Ages 5-7)
Description: The impact on quality of life (QOL) was measured by a general pediatric health questionnaire. Versions were self-administered & answered by participants' parents. Questionnaire consists of 23 items using a 3-point scale: from 0 (not at all), 2 (sometimes), 4 (a lot). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored. Total score is sum of all the items over the number of items answered on all the scales. Higher scores indicate a better health related QOL.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: The ITT population included all randomized participants who received >= 1 dose after commencement of treatment. At baseline (visit 2), 52 randomized participants were between 5 and 7 years old, 28 participants in MFNS & 24 subjects in Placebo group. Questionnaire was answered in accordance with the actual age of each participant at each visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 28 | 24
Score on a scale
  Visit 2 (n= 28 MFNS, n=24 Placebo) | 78.14 (15.74) | 79.03 (11.35)
  Visit 3 (n=28 MFNS, n= 23 Placebo) | 81.56 (13.64) | 84.07 (12.26)
  Visit 4 (n=28 MFNS, n=22 Placebo) | 83.54 (13.63) | 82.71 (13.52)

19. Secondary Outcome: Quality of Life Questionnaire (PedsQL) Total Score (Ages 8-12)
Description: The impact on quality of life (QOL) was measured by a general pediatric health questionnaire. Versions were self-administered & answered by participants' parents. This modular instrument consists of 23 items using a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored. Total score is sum of all the items over the number of items answered on all the scales. Higher scores indicate a better health related QOL.
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: The ITT population included all randomized participants who received >= 1 dose after commencement of treatment. At baseline (visit 2), 28 randomized participants were between 8-12 years old, 15 participants in MFNS & 13 participants in Placebo group. Questionnaire was answered in accordance with the actual age of each participant at each visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 15 | 18
Score on a scale
  Visit 2 (n= 15 MFNS, n=13 Placebo) | 76.014 (10.266) | 76.839 (10.828)
  Visit 3 (n=15 MFNS, n= 14 Placebo) | 82.971 (15.054) | 84.006 (14.033)
  Visit 4 (n=15 MFNS, n=13 Placebo) | 85.725 (12.033) | 83.946 (10.023)

20. Secondary Outcome: Obstructive Sleep Apnea-18 (OSA-18) Questionnaire Total Score
Description: 18 items of the survey were graded on a 7-point ordinal scale. Caregivers were asked to describe how often in the last 4 weeks had the child exhibited specific symptoms according to the following scale: 1: none of the time; 2: hardly any of the time; 3: a little of the time; 4: some of the time; 5: a good bit of the time; 6: most of the time; 7: all of the time. All scores were summed (total score: 18-126).
  Grading was as follows:
  * Scores < 60 suggest a slight impact on health related quality of life (HRQL)
  * Scores 60-80 suggest a moderate impact
  * Scores over 80 suggest a great impact
Time Frame: Baseline (Visit 2), Week 4 (Visit 3), Week 8 (Visit 4)
Population: A total of 132 subjects were included in the ITT population. The ITT population included all randomized participants who received >=1 dose after commencement of treatment. Data summarized in terms of the number of participants providing data at the relevant time point.
  1 participant in Placebo group did not answer this questionnaire at baseline.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray (MFNS) | Placebo Nasal Spray
Number analyzed (Participants) | 66 | 66
Score on a scale
  Visit 2 (n=66 MFNS, n=65 Placebo) | 62.742 (19.951) | 60.169 (19.123)
  Visit 3 (n=65 MFNS, n= 65 Placebo) | 47.138 (18.806) | 48.769 (18.748)
  Visit 4 (n=62 MFNS, n= 59 Placebo) | 42.742 (17.880) | 43.068 (18.870)

ADVERSE EVENTS:
Time Frame: Up to Week 24
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 2/66 | 3/66
Other Adverse Events (participants affected / at risk) | 18/66 | 17/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=66) | Placebo Nasal Spray (N=66)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=66) | Placebo Nasal Spray (N=66)
Pyrexia (General disorders) | 5 (10) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Pharyngitis (Infections and infestations) | 4 (7) | 3 (4)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 4 (6)
Sinusitis (Infections and infestations) | 4 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (14)

LIMITATIONS AND CAVEATS:
The results of this study as presented are drawn from the clinical study report and should be reviewed with caution as there were inaccuracies in the database resulting from medication errors in some participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees not to publish or publicly present any interim results of the Study without prior written consent of the SPONSOR. The Principal Investigator further agrees to provide thirty (30) days written notice to the SPONSOR prior to submission for publication or presentation to permit the SPONSOR to review copies of abstracts or manuscripts for publication which report any results of the Study.